CLINICAL TRIAL: NCT00984217
Title: Phase II Trial of Postoperative Radiotherapy and Panitumumab in High-risk Salivary Gland Malignancies
Brief Title: Trial of Radiotherapy and Panitumumab in Salivary Gland Malignancies
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Decided not to pursue at UPCI
Sponsor: University of Pittsburgh (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-112
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Adenoma, Pleomorphic; Mixed Salivary Gland Tumor; Salivary Gland Tumor, Mixed; Syringoma, Chondroid
Keywords: panitumumab; salivary gland malignancies; radiotherapy
MeSH Terms: conditions — Adenoma, Pleomorphic | interventions — Radiation; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Panitumumab (Experimental): Panitumumab 2.5 mg/Kg IV, weekly during radiation (total of 6-8 doses).
  Interventions: Radiation: Radiation; Drug: Panitumumab

INTERVENTIONS:
Radiation: Radiation — Radiation 64-70Gy (2.0 Gy/day, 5 days/week)
Drug: Panitumumab — 2.5 mg/Kg IV, weekly during RT. 6-7 weeks

SUMMARY:
Standard therapy for high-risk or locally advanced salivary gland malignancies is surgery followed by postoperative radiation therapy. Retrospective studies have shown the superiority of combined modality therapy compared to surgery alone for patients with advanced T or N stage. Despite the addition of postoperative radiation therapy, the five-year survival for locally advanced salivary gland malignancies is poor (less than 60%). In salivary gland malignancies, the epidermal growth factor receptor (EGFR) is expressed in 25-85%; in certain histological types, like salivary duct carcinomas, the expression is higher. EGFR is a promising target of anticancer therapy. In squamous cell carcinoma of the head and neck, a phase III trial utilizing cetuximab added to radiation therapy improved both locoregional control and overall survival compared to radiation alone. Panitumumab is a novel, human, IgG2 EGFR monoclonal antibody that may be better tolerated and more efficacious than cetuximab. Here, the investigators suggest that the addition of panitumumab to standard radiotherapy in locally-advanced salivary gland malignancies will improve recurrence-free survival (RFS).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically determined salivary gland cancer of the major or minor salivary glands of the head and neck (any histology) status post potentially curative surgical resection with no macroscopic residual disease. Patients should have AJCC 6th edition stage III with:

  1. extracapsular extension,
  2. perineural invasion,
  3. positive surgical margins or
  4. high grade histology (i.e., high grade mucoepidermoid carcinoma, adenocarcinoma except basal cell adenocarcinoma, salivary duct carcinoma, squamous cell carcinoma, or adenoid cystic carcinoma) or stage IVA or IVB.
* No distant metastasis.
* No prior chemotherapy, biologic/targeted therapy (including any prior therapy which specifically and directly targets the EGFR pathway), or radiotherapy for head and neck cancer.
* No more than 10 weeks (minimum of 3 weeks) should elapse between surgery and treatment on study.
* ECOG performance status of 0-2
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count: Greater than or equal to 1500/uL
  * Platelets: Greater than or equal to 100,000/uL
  * Hemoglobin: Greater than or equal to 10g/dL
  * Total bilirubin: < 1.5x normal institutional limits
  * Creatinine clearance: > 45 mL/min
  * Magnesium level: > lower limit normal
* No prior invasive malignancy unless the disease-free survival is 3 years or more.
* Age greater than or equal to 18 years
* Pregnant or breast-feeding women are excluded (see exclusion criteria).
* Informed consent must be obtained from all patients prior to beginning therapy. Patients should have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction. All patients will have a baseline EKG. If abnormalities consistent with active coronary artery disease are detected, the patient will be referred to a cardiologist for appropriate evaluation and management prior to treatment on study.
* Patients may not be receiving any other investigational agents.
* No history of prior malignancy, with the exception of basal carcinoma of the skin or in situ cervical cancer, or malignancy that has been treated with a curative intent with a 3-year disease-free survival.
* Pregnant women are excluded from this study because chemotherapy and radiation therapy have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with chemotherapy, breastfeeding should be discontinued if the mother is treated with chemotherapy. Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control.

  * All WOCBP MUST have a negative urine pregnancy test at baseline, or within 7 days prior to receiving investigational product. The minimum sensitivity of the pregnancy test must be 25 IU/L or equivalent units of HCG. If the urine pregnancy test is positive, a serum pregnancy test will then be performed to confirm the result. In the event that both the urine and serum pregnancy tests are positive, the subject must not receive investigational product and must not be enrolled in the study.
  * In addition, all WOCBP should be instructed to contact the Investigator immediately if they suspect they might be pregnant (e.g., missed or late menstrual period) at any time during study participation.
  * The Investigator must immediately notify Amgen in the event of a confirmed pregnancy in a patient participating in the study.
* Prior severe infusion reaction to a human monoclonal antibody.
* Prior radiotherapy, chemotherapy or EGFR inhibitor for head and neck cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the recurrence-free survival of advanced salivary gland cancer patients undergoing postoperative chemoradiotherapy with panitumumab compared to historical control data | 3 years

SECONDARY OUTCOMES:
To evaluate the overall survival, local recurrence-free survival, distant recurrence-free survival and toxicities. | 3 years
To correlate efficacy parameters with a) EGFR and downstream pathway activation, b) FcyR polymorphisms, and c) serum cytokine profiles. | 3 years
To collect tumor tissue from pretreatment biopsies for cytokine/chemokine and immune biomarker studies on tumor tissue. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael K. Gibson, MD, Principal Investigator — University of Pittsburgh
Locations (27):
- United States (27):
  - UPMC Cancer Center - Teramana Cancer Center - Steubenville, Steubenville, Ohio
  - UPMC Cancer Center - Beaver, Beaver, Pennsylvania
  - UPMC Cancer Center - Clairton, Clairton, Pennsylvania
  - UPMC Cancer Center - Arnold Palmer Pavilion - Greensburg, Greensburg, Pennsylvania
  - UPMC Cancer Center - Oakbrook Commons - Greensburg, Greensburg, Pennsylvania
  - UPMC Cancer Center - Oakbrook Commons, Greensburg, Pennsylvania
  - UPMC Cancer Center -Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Cancer Center - Indiana, Indiana, Pennsylvania
  - UPMC Cancer Center - John P. Murtha Pavilion - Johnstown, Johnstown, Pennsylvania
  - UPMC Cancer Center - McKeesport, McKeesport, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Cancer Center - Sewickley Medical Oncology/Hematology Group, Moon Township, Pennsylvania
  - UPMC Cancer Center -Mt. Pleasant, Mount Pleasant, Pennsylvania
  - UPMC Cancer Center - New Castle, New Castle, Pennsylvania
  - UPMC Presbyterian -Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC Cancer Center - St. Margaret's, Pittsburgh, Pennsylvania
  - UPMC Cancer Center -Delafield Rd., Pittsburgh, Pennsylvania
  - Hillman Cancer Center: University of Pittsburgh Cancer Institute / UPMC Department of Radiology, Pittsburgh, Pennsylvania
  - UPMC Cancer Center -UPMC Shadyside, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - UPMC Cancer Center - Passavant, Pittsburgh, Pennsylvania
  - UPMC Cancer Center - Upper St. Clair, Pittsburgh, Pennsylvania
  - UPMC Cancer Center -Drake, Pittsburgh, Pennsylvania
  - UPMC Cancer Center -UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center - Uniontown, Uniontown, Pennsylvania
  - UPMC Cancer Center - Washington, Washington, Pennsylvania
  - UPMC Cancer Center - North Hills, Wexford, Pennsylvania